CLINICAL TRIAL: NCT05788276
Title: Can Dapagliflozin Preserve Structure and Function in Transplanted Kidneys?
Acronym: DEAKTransplant
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: St. Olavs Hospital (Other); University Hospital of North Norway (Other); Haukeland University Hospital (Other)
Responsible Party: Principal Investigator, Trond Jenssen, Chef Physician at Department of Organ Transplantation, Professor of Nephrology, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2022/426076
Record Dates: First submitted 2023-01-26; First posted 2023-03-28 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Kidney Transplant; Complications; Kidney Transplant Failure; Renal Failure
Keywords: Kidney; Transplantation; SGLT2; Renal function
MeSH Terms: conditions — Renal Insufficiency | interventions — dapagliflozin; Exercise

STUDY DESIGN:
Intervention Model Description: Randomized, Double blinded, placebo controlled interventional study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active treatment (Active Comparator): 165 patients
  Interventions: Drug: Dapagliflozin 10mg Tab
- Control group (Placebo Comparator): 165 patients
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dapagliflozin 10mg Tab — Dapagliflozin active tablets
  Other Names: Active
  Arms: Active treatment
Drug: Placebo — Matched placebo tablets
  Arms: Control group

SUMMARY:
The goal of this clinical trial is to look at the effect of SGLT2 (Sodium glucose transporter 2) inhibition in patients receiving a kidney-transplant 6 weeks earlier at Oslo University hospital. Rikshospitalet. Investigators will search for answers along three pathways: Can SGLT2 inhibitor 1) preserve glomerular filtration rate (GFR), 2) reduce interstitial fibrosis in the kidney, and 3) favorably improve metabolic risk factors for graft failure such as visceral obesity, glucose intolerance and high blood pressure? The participants (N=330) will be randomized to either dapagliflozin 10 mg or placebo o.d. in a blinded fashion. Researchers will than use kidney transplant biopsies, measured GFR, blood pressure sampling, glucose tolerance test (OGTT), dual-energy X-ray absorptiometry (DXA scan) and estimated GFR from the two groups in comparison, to evaluate the effect treatment. The participants will be followed for a total of 3 years.

DETAILED DESCRIPTION:
This is a randomized, placebo-controlled trial with dapagliflozin 10 mg vs. placebo o.d. in kidney transplant patients. The patients are randomized 1:1 to active: placebo treatment 6 weeks after transplantation and followed for a total of 150 weeks (156 weeks post-transplant).

Before treatment initiation (6 weeks after transplantation) the following investigations will be performed;

1. Estimated GFR: Assessed using the Modification of Diet in Renal Disease 4 (MDRD-4) formula and is presented as mL/min/1.73 m2. Plasma creatinine concentrations are to be analyzed at the Department of Medical Biochemistry where the patient is followed and is presented as mmol/L. (Estimated GFR will be calculated from at least 4 plasma creatinine measurements per year).
2. Blood sample: Measured variables include plasma creatinine, hemoglobin, hematocrit, sodium, potassium, magnesium and uric acid.
3. Kidney tissue analyses: a.) Light microscopical evaluation in formalin-fixed and paraffin-embedded (FFPE) kidney graft biopsies: Semi-quantitative estimation of percent graft fibrosis in the renal cortex according to the Banff classification, percent interstitial fibrosis and percent inflammation outside fibrotic scars. b.) Immunohistochemistry: Graft samples will be deparaffinized and boiled in antigen retrieval solution and then exposed to primary antibodies against collagen and extracellular matrix markers, e.g. periostin, tenascin and picrosirius red. In addition, p16INKa, a marker of premature aging, and endothelial markers to evaluate capillary density will be used.

   c.) Samples will be digitally scanned to perform digital morphometric evaluation using the softwares 3D Histech, Analysis Pro and QuPath. Areas not of interest (renal medulla, scar tissue, capsule or subscapular areas), poor quality scans and artefacts will be excluded. Digital software will also be used to estimate glomerular volume and mesangial volume fraction using QuPath. All evaluations will be performed by investigators blinded for the study participants' identity and clinical data. This is an explorative study, and no power estimate is available.

   d.) The investigators will also perform molecular analyses, mRNA and proteomics in a subsample (n=25 in intervention, n=25 in control group, matched for age, gender and eGFR as appropriate) at the same two time-points as described above (altogether n=100 biopsies processed for RNA sequencing and proteomics), using standard bulk mRNA/miRNA sequencing and proteomics of whole sections from 'RNA later' kidney graft biopsies (Genomics and Proteomics Core Facilities, UiO). The investigators will also perform bioinformatic analyses focusing on fibrosis.
4. Oral glucose tolerance test (OGTT): Will be performed in persons not on glucose-lowering treatment by ingestion of 75 g glucose dissolved in water (or 1 g/kg if body weight is <75 kg). Blood samples for measurements of glucose, insulin and C-peptide are collected at 0, 30 and 120 min, respectively. Glucose tolerance is assessed by the 2-h glucose value, while first phase insulin release is primarily reflected by the 30 min insulin value which is included in the Stumvoll equation which measures both first and second phase insulin release. Insulin sensitivity will be assessed by the Matsuda equation.
5. Protein/creatinine ratio: Will be assessed at the Department of Medical Biochemistry where the patient is followed. Open urinary stix is not considered appropriate, partly due to the risk of unblinding in case of glucosuria detection by a combined stix. (Protein/ creatinine ratio will be collected from at least 4 urine sample measurements per year)
6. Blood Pressure: Will be assessed as both systolic and diastolic measure, and measurements are performed according to standard procedures (measured in mmHg ). The same standard will be followed for blood pressure measurements at the local hospitals.
7. Metabolomics: Urine and serum will be sent on dry ice in larger batches. LC-MS methodology will be used for the analysis, using a commercial kit (Biocrates). ELISA methodology will in addition be used in case verification analyses are necessary. This exploratory analysis will focus on markers for fibrosis, inflammation and secretion function in the kidney tubuli.

   After 2 weeks the patients will go through repeated blood sampling and blood pressure measurements, followed by the following procedures;
8. Measured GFR: Assessed at the Laboratory for Renal Physiology, by the iohexol serum clearance method utilizing the Bayesian estimate 4-point method. Serum samples are to be obtained 10 min, 30 min, 2 h and 5 h after administration of 5 mL Omnipaque (300 mg I/mL). measured GFR (Iohexol serum clearance) and DXA assessed body composition (subcutaneous and visceral fat percentage of total fat mass) is assessed, after 72 weeks of treatment all investigations/biobanking performed before and after 2 weeks are repeated. Then, after 150 weeks, the final visit is performed, including blood pressure measurements and the urinary protein/creatinine ratio and clinical chemistry determinations.
9. DXA scan: Total body composition will be determined by a narrow fan-beam Lunar Prodigy Densitometer (GE Healthcare) and all the scans will be analysed using enCORER software version 14.10 (GE Medical Systems, Lunar Corp., Madison, WI). The automated software is capable of discriminating subcutaneus adipose tissue (SAT) and visceral adipose tissue (VAT) within android region of interest (ROI). In vivo, short-term coefficients of variation for total body tissue and lean and fat mass are 0.1%, 0.8%, and 2.5%. The VAT short-term repeat measurement error coefficient of variation is 9.8% DXA-derived VAT was previously validated against CT, the standard method for the quantitative assessment of intra abdominal adipose tissue.

At week 78 patients will go through repeated analyses of the tests listed above. They will also go through 24 hour blood pressure tests 8 weeks, 72 weeks and 150 weeks after randomization.

Throughout the study all plasma creatinine and urinary protein/creatinine ratios will be included in the study clinical research form (CRF). Safety measures will also be included. Measured GFR will measure the chronic GFR slope, while estimated GFR will assess the total GFR slope (both the early dip and the chronic slope of GFR). Furthermore, after the final study visit, which represents150 weeks of blinded treatment, all patients will be allowed further open treatment with SGLT2-inhibitors to the discretion of the treating physician and the patient. Furthermore, eGFR slope, graft loss and cardiovascular events will be followed based on annual data from the Norwegian Renal Registry for up to 10 years after transplantation.

For a more detailed description of primary and secondary objectives and endpoints see bellow.

ELIGIBILITY:
Inclusion Criteria:

* Renal transplant recipients transplanted 6 weeks earlier at Oslo University hospital (OUH) Rikshospitalet.
* Age 18-75 years.
* Able to comply with the medical treatment on their own.
* Calcineurin inhibitor trough concentrations in accordance with individual therapeutic range and standard dose prednisolone and mycophenolate mofetil over the last 2 weeks.
* Estimated GFR ≥25 mL/min/1.73 m2.

Exclusion Criteria:

* Type 1 diabetes
* Rejection episodes of the kidney graft prior to randomization.
* Ongoing infectious disease or intermittent causes affecting renal function, e.g., obstructive lymphocele.
* Malnutrition.
* Urosepsis less than 1 year prior to randomization.
* Participants with a known hypersensitivity to dapagliflozin or any of the excipients of the product.
* For women only - currently pregnant

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330 (Estimated)
Dates: Start 2023-05-02 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Effect of Dapagliflozin on the GFR slope in renal transplant patients (Main study) | From before randomization to 3 years after transplantation.
  1. Difference in eGFR slope between groups.

SECONDARY OUTCOMES:
The effect of Dapagliflozin on renal and metabolic conditions between groups (Main study) | From before randomization to 3 years after transplantation
  1. Change in measured GFR (iohexol serum clearance)
  2. Change in mean arterial blood pressure in mmHg
  3. Change of DXA-measured visceral fat (grams)
  4. Change in hematocrit (%)
  5. Change in two hour blood glucose measured by an oral glucose tolerance test in patients without diabetes (mmol/L).
  6. Change in urine protein/creatinine ratio (mg/mmol)
Changes in renal graft fibrosis and proteomic markers with SGLT2 inhibition between groups (Sub-study - the 140 first included patients). | From before randomization to 3 years after transplantation
  1. Change in inflammation score
  2. Change in fibrosis score
  3. Change in kidney graft mRNA score
  4. Change in proteomic score

CONTACTS AND LOCATIONS:
Overall Officials: Trond Geir Jenssen, MD, Principal Investigator — Oslo University Hospital
Locations (1):
- Oslo University Hospital, Oslo, Oslo County, Norway

IPD SHARING:
Plan to Share IPD: No
So far undecided, but application to regional ethics committee (REC) is possible if it is desirable.